CLINICAL TRIAL: NCT03537261
Title: Crisis Prevention Institute (CPI) Verbal and Physical Management Training for Parents of Children With ASD (P-CPI)
Brief Title: CPI Training for Parents of Children With ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Crisis Prevention Institute (Other)
Responsible Party: Principal Investigator, Lisa A. Nowinski, PhD, Director, Neuropsychology Training, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018P000119
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Results first posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Autism Spectrum Disorder
Keywords: Parent Training; Aggressive Behavior
MeSH Terms: conditions — Autism Spectrum Disorder; Aggression | interventions — cyclopropapyrroloindole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPI-Parent Training (Experimental): Will receive one-day (6-hour) training in P-CPI including the use of nonverbal, paraverbal, verbal, and physical intervention techniques.
  Interventions: Behavioral: Parent-based Crisis Prevention Institute (CPI) physical management training program (P-CPI)
- Waitlist Control (No Intervention): Will not receive active P-CPI training during the experimental treatment interval.
  NOTE: The waitlist group will be offered the P-CPI training session after the treatment group completes their follow-up measures.

INTERVENTIONS:
Behavioral: Parent-based Crisis Prevention Institute (CPI) physical management training program (P-CPI) — Parents of children with ASD will be randomly assigned to the 6-hour P-CPI group training session, which includes nonverbal, paraverbal, verbal, and physical intervention techniques. Baseline measures will be administered on the day of training and follow-up measures at 2-week, 1-month, 2-month, and 3-month post baseline. The treatment group will also participate in an in-person follow-up group qualitative interview.
  Other Names: (P-CPI)
  Arms: CPI-Parent Training

SUMMARY:
The purpose of this 24-week study is to determine whether the "Parent-based Crisis Prevention Institute (CPI) physical management training program" (i.e., P-CPI) is effective in increasing self-efficacy in parents of children with autism spectrum disorder (ASD).

DETAILED DESCRIPTION:
Parents of children with ASD deal with more stress, especially if their child demonstrates self-injurious and aggressive behavior. The purpose of this study is to evaluate whether "Parent-based Crisis Prevention Institute (CPI) physical management training program" (i.e., P-CPI) for parents of children with ASD helps alleviate some of this stress and increase parental self-efficacy, physical management competency, and overall quality of life.

Participants who meet criteria will be randomly assigned to either the treatment group or the waitlist control group. Participants assigned to the treatment group will be invited to a 6-hour P-CPI group training session. This parent-based training in CPI's Nonviolent Crisis Intervention® will include nonverbal, paraverbal, verbal, and physical intervention techniques. Participants assigned to the waitlist group will be encouraged to continue their existing medical support, or services, as they typically would. The waitlist group will be invited to participate in the P-CPI training at the conclusion of the post-assessment period.

Baseline measures will be on the day of training for the treatment group and within five days of the P-CPI training for the waitlist group. Follow-up measures will be at 2-week, and 1, 2, and 3- month post-baseline. The treatment group will also participate in a follow-up group interview.

ELIGIBILITY:
Inclusion Criteria:

* Each subject must be an adult caregiver/parent of a Lurie Center for Autism patient with 'patient' defined as having at minimum one visit/contact per year with any Lurie Center for Autism clinician. The patient (child):

  * May be male or female.
  * Must be from 5-12 years of age (inclusive).
  * Must live at home.
  * May have any IQ.
  * Must have an ASD diagnosis per the DSM-5 checklist confirmed by expert clinician at enrollment.
  * Must have a symptom severity score of 18 or greater on the ABC Irritability subscale confirmed by expert clinician at enrollment.
* The subject may have any primary language but must be comfortable speaking and reading English without translation.
* The subject must be the self-identified primary caregiver of the Lurie Center for Autism patient.
* The subject must be recommended by a Lurie Center for Autism clinician.
* The subject must be able to attend in person the maximum the training session on the specified date/time/location.
* The subject must be willing to complete the assessment measures.
* Only one subject per family may participate.

Exclusion Criteria:

* The subject must not have any self-identified physical limitations or disabilities that prevent use of physical intervention techniques.
* The patient (child) of the subject must not have any compromising neurological disorders (i.e., CP, active seizures).
* The patient should not have the addition of non-drug treatment (including ABA and parent-training) for 4 weeks prior to intervention

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Nowinski, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Lurie Center for Autism, Lexington, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant withdrew consent prior to randomization.
Period: Overall Study
Arm/Group | CPI-Parent Training | Waitlist Control
Started | 41 | 39
Completed Baseline Assessment | 35 (One participant did not attend the CPI-Parent training but remained in the study.) | 28
Completed | 33 (One participant did not attend the CPI-Parent training but remained in the study.) | 27
Not Completed | 8 | 12
Not completed — Lost to Follow-up | 4 | 5
Not completed — Withdrawal by Subject | 4 | 6
Not completed — Did not return study questionnaires | 0 | 1

BASELINE CHARACTERISTICS:
Population: Six participants assigned to CPI-Parent training and 11 participants assigned to waitlist discontinued study participation prior to baseline assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | CPI-Parent Training | Waitlist Control | Total
Number analyzed (Participants) | 35 | 28 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 28 | 63
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 25 | 57
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 34 | 26 | 60
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 31 | 27 | 58
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 28 | 63
Child Adjustment and Parent Efficacy Scale-Developmental Disability Self-Efficacy Scale Total Score [Mean (Standard Deviation); unit: units on a scale] — The CAPES-DD self-efficacy scale is a 16-item brief outcome measure in the evaluation of individual parenting interventions that measures parents' self-efficacy in managing specific child behavior problems. Instructions were modified to ask about the previous two weeks instead of the previous four weeks. The range of possible scores is 16-160, with higher scores corresponding to greater parental self-efficacy.
  units on a scale | 111.3 (21.8) | 101.3 (17.8) | 106.8 (20.6)
Parent Stress Index - Short Form Total Score [Mean (Standard Deviation); unit: units on a scale] — The PSI-SF is a self-report measure of severity and domain of parenting stress which includes 36 items rated on a 5-point, Likert scale. The range of possible values for the total stress raw score is 36-180, with higher scores corresponding to greater levels of parental stress.
  units on a scale | 115.0 (19.4) | 117.6 (21.0) | 116.2 (20.0)
Family Quality of Life Scale Total Score [Mean (Standard Deviation); unit: units on a scale] — The FQOL scale is a 25-item measure assessing families' perceptions of their satisfaction with different aspects of family quality of life. It assesses five domains: family interaction, parenting, general resources, health and safety, and support for persons with disabilities. Instructions were modified to ask about the previous two weeks instead of the previous 12 months. The range of possible values for the FQOL total score is 25-125, with higher scores corresponding to better quality of life.
  units on a scale | 93.3 (11.8) | 90.5 (13.9) | 92.1 (12.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Child Adjustment and Parent Efficacy Scale-Developmental Disability Self-Efficacy Scale Total Score
Description: The CAPES-DD self-efficacy scale is a 16-item brief outcome measure in the evaluation of individual parenting interventions that measures parents' self-efficacy in managing specific child behavior problems. Instructions were modified to ask about the previous two weeks instead of the previous four weeks. The range of possible scores is 16-160, with higher scores corresponding to greater parental self-efficacy and a positive change indicating improvement from baseline. Mean changes were estimated using repeated measures linear regression controlling for score at screening visit.
Time Frame: Baseline and 2-weeks
Population: All 35 participants assigned to P-CPI training and 28 participants assigned to waitlist who completed the baseline assessment contributed at least one CAPES-DD self-efficacy total score to the analysis. Five of these participants contributed only one score: two assigned to P-CPI training and one assigned to waitlist who discontinued study participation between baseline and two weeks, and one at baseline and one at two weeks assigned to P-CPI training who provided incomplete CAPES-DD data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | CPI-Parent Training | Waitlist Control
Number analyzed (Participants) | 35 | 28
units on a scale | 8.3 [3.3 to 13.3] | 2.5 [-2.9 to 7.8]
Statistical Analysis 1: Comparison: CPI-Parent Training vs Waitlist Control; Test type: Superiority; p = 0.11, Regression, Linear; Repeated measures linear regression controlling for score at screening visit; Mean Difference (Net) = 5.8, 95% CI 2-sided [-1.4 to 13.1] — (P-CPI training change) - (waitlist change)

2. Secondary Outcome: Change in the Parent Stress Index - Short Form Total Score
Description: The PSI-SF is a self-report measure of severity and domain of parenting stress which includes 36 items rated on a 5-point, Likert scale. The range of possible values for the total stress raw score is 36-180, with higher scores corresponding to greater levels of parental stress and negative change corresponding to reduced levels of parental stress. Mean changes were estimated using repeated measures linear regression controlling for score at screening visit.
Time Frame: Baseline and 2-weeks
Population: All 35 participants assigned to P-CPI training and 28 participants assigned to waitlist who completed the baseline assessment contributed at least one PSI-SF total score to the analysis. Five of these participants contributed only one score: two assigned to P-CPI training and one assigned to waitlist who discontinued study participation between baseline and two weeks, and two at two weeks assigned to P-CPI training who provided incomplete PSI-SF data or did not complete the scale.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | CPI-Parent Training | Waitlist Control
Number analyzed (Participants) | 35 | 28
units on a scale | -2.7 [-6.3 to 0.8] | -0.5 [-4.4 to 3.3]
Statistical Analysis 1: Comparison: CPI-Parent Training vs Waitlist Control; Test type: Superiority; p = 0.40, Regression, Linear; Repeated measures linear regression controlling for score at screening visit; Mean Difference (Net) = -2.2, 95% CI 2-sided [-7.4 to 3.0] — (P-CPI training change) - (waitlist change)

3. Secondary Outcome: Change in the Family Quality of Life Scale Total Score
Description: The FQOL is a 25-item measure assessing families' perceptions of their satisfaction with different aspects of family quality of life. It assesses five domains: family interaction, parenting, general resources, health and safety, and support for persons with disabilities. Instructions were modified to ask about the previous two weeks instead of the previous 12 months. The range of possible values for the FQOL total score is 25-125, with higher scores corresponding to better quality of life and positive change corresponding to improved quality of life. Mean changes were estimated using repeated measures linear regression controlling for score at screening visit.
Time Frame: Baseline and 2-weeks
Population: All 35 participants assigned to P-CPI training and 28 participants assigned to waitlist who completed the baseline assessment contributed at least one FQOL total score to the analysis. Four of these participants contributed only one score: two assigned to P-CPI training and one assigned to waitlist who discontinued study participation between baseline and two weeks, and one at baseline assigned to waitlist who provided incomplete FQOL data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | CPI-Parent Training | Waitlist Control
Number analyzed (Participants) | 35 | 28
units on a scale | 1.9 [-0.5 to 4.3] | 1.3 [-1.4 to 4.0]
Statistical Analysis 1: Comparison: CPI-Parent Training vs Waitlist Control; Test type: Superiority; p = 0.72, Regression, Linear; Repeated measures linear regression controlling for score at screening visit; Mean Difference (Net) = 0.6, 95% CI 2-sided [-2.9 to 4.2] — (P-CPI training change) - (waitlist change)

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Events determined by the Principal Investigator (PI) to be unanticipated problems involving risks to participants or others were to be reported by the PI according to the Partners Human Research Committee's reporting policies.
Arm/Group | CPI-Parent Training | Waitlist Control
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/28
Other Adverse Events (participants affected / at risk) | 0/35 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT03537261/Prot_SAP_000.pdf